CLINICAL TRIAL: NCT03523910
Title: Right Ventricular Pulmonary Vascular Interaction in Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-1526; 1R01HL105598-01A1 (NIH)
Record Dates: First submitted 2018-02-26; First posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Single center, open label, single-arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient (Experimental): A research MRI scan with exercise will be obtained in conjunction with standard of care cardiopulmonary testing.
  Interventions: Device: Magnetic Resonance Imaging (MRI) with exercise

INTERVENTIONS:
Device: Magnetic Resonance Imaging (MRI) with exercise — MRI scan with a novel exercise device.
  Other Names: MRI

SUMMARY:
The goals of this study were two-fold. First, the attempt to quantify the relationships between pulmonary arterial stiffness, right ventricular function and the efficiency of ventricular-vascular interactions in patients with pulmonary arterial hypertension (PAH). Second, the attempt to quantify the effects of exercise on pulmonary arterial stiffness, pulmonary vascular resistance, right ventricular function and the efficiency of ventricular-vascular interactions in patients with PAH.

DETAILED DESCRIPTION:
The goals of this study are to quantify right ventricular-pulmonary vascular interactions in different types of PAH, to determine the temporal changes in these interactions with PAH progression and to quantify the effects of exercise on right ventricular function. The inclusion of the subpopulation of PAH patients with systemic sclerosis (SSc) was a result of the anticipation that this group has worse arterial stiffening than other groups, and consequently more inefficient right ventricular-pulmonary vascular interactions, which account for their worse prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of pulmonary arterial hypertension or a subtype
2. Referred for right heart catheterization
3. Age between 18 and 80 years
4. New York Heart Association (NYHA) functional class I, II, or III

Exclusion Criteria:

1. Recent syncope (within 1 year)
2. Severe skeletal or muscle abnormalities prohibiting exercise
3. Mixed etiology pulmonary arterial hypertension
4. Severe lung disease

   1. Test results indicating severe obstruction
   2. Total lung capacity < 60%
5. Pregnancy or breastfeeding
6. NYHA class IV patient
7. Contraindications to magnetic resonance imaging
8. Kidney dysfunction as determined by an estimated glomerular filtration rate (eGFR) of < 30 mL/min/1.73m2
9. Contraindication to gadolinium

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-04-25 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2017-02-13 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to comprehensively quantify right ventricular and pulmonary vascular function at rest and with exercise using magnetic resonance imaging. | Up to 24 months
  The hypotheses will be tested by comprehensively quantifying ventricular and vascular function in subjects with idiopathic pulmonary arterial hypertension, systemic sclerosis pulmonary arterial hypertension, and chronic thromboembolic pulmonary hypertension, using investigational magnetic resonance angiography techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Francois, MD, Principal Investigator — University of Wisconsin, Madison

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Macdonald JA, Franҫois CJ, Forouzan O, Chesler NC, Wieben O. MRI assessment of aortic flow in patients with pulmonary arterial hypertension in response to exercise. BMC Med Imaging. 2018 Dec 22;18(1):55. doi: 10.1186/s12880-018-0298-9. PMID 30577768